CLINICAL TRIAL: NCT05058248
Title: "Evaluation of a Locoregional Anesthesia Protocol by Pudendal Block in Reconstructive Surgery Clitoral " Pudendal Block in Clitoral Surgery (Pain REparation CLItoris)
Brief Title: Evaluation of a Locoregional Anesthesia Protocol by Pudendal Block in Reconstructive Surgery Clitoral
Acronym: DORECLI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Raincy Montfermeil Hospital Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHIM -RIPH2-001
Record Dates: First submitted 2021-09-13; First posted 2021-09-27 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2021-09

CONDITIONS: Reduction in Pain Within 24 Hours of Surgery
Keywords: excision; Reconstructive surgery of the clitoris; sexual health; chronic pain,; The pudendal block nerve endings.; postoperative pain in clitoral surgery
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Prospective non-randomized study comparing the group of patients who received general anesthesia and pudendal block in a historical cohort of patients treated by the standard establishment protocol, that is to say under general anesthesia without locoregional anesthesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pudendal block (Active Comparator): Ultrasound-guided bilateral pudendal block at the start of surgery, in gynecological position: injection of 15 mL of 0.475% Naropein in each ischiorectal fossa.
  Interventions: Procedure: pudendal block
- the standard method (Other): Operated and anesthetized patients according to the standard method within the department
  Interventions: Procedure: pudendal block

INTERVENTIONS:
Procedure: pudendal block — general anesthesia with an intravenous analgesic protocol then oral without anesthesia regional loco
  Other Names: standard method

SUMMARY:
Reconstructive surgery of the clitoris is part of the care offered during a process of care of women victims of MSF. It consists in reconstituting a clitoral neogland after removal of the vulvar excisional scar and recovery of the remaining clitoris. Studies that have monitoring the implementation of this surgery show that it improves the well-being of the patients, brings benefits anatomically, sexual health, personal development, and in the long term decreases chronic pain.

Currently the standard method used in the usual care of the patient is: general anesthesia with an intravenous analgesic protocol then oral without anesthesia regional loco The pudendal block that the investigators want to evaluate in this research, is a technique that has made proven in several types of surgery, associated with very few complications and easily reproducible.

DETAILED DESCRIPTION:
Reconstructive surgery of the clitoris is part of the care offered during a process of care of women victims of MSF. It consists in reconstituting a clitoral neogland after removal of the vulvar excisional scar and recovery of the remaining clitoris. Studies that have monitoring the implementation of this surgery show that it improves the well-being of the patients, brings benefits anatomically, sexual health, personal development, and in the long term decreases chronic pain. Currently the standard method used in the usual care of the patient is: general anesthesia with an intravenous analgesic protocol then oral without anesthesia regional loco The pudendal block that the investigators want to evaluate in this research, is a technique that has made proven in several types of surgery, associated with very few complications and easily reproducible. The human clitoris is the most sensitive organ in the human body, with over 8000 endings nervous. All these endings come from the pudendal nerve, itself most often of nerve roots S3. The main hypothesis is that a bilateral anesthetic block of this nerve would reduce postoperative pain in clitoral surgery

ELIGIBILITY:
Inclusion Criteria:

* Major patient,
* With the indication of a clitoral repair surgery
* Having expressed their free and informed written consent
* Affiliated with a social security scheme

Exclusion Criteria:

- Contraindication to the pudendal block technique: notably :

* blood crass disorder
* allergy to Naropein
* infection at the injection site - Poor understanding of the interest of the practice proposed experimental

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
decrease in the mean of the self-reported pain scores in the first 24 hours | 24 hours
  decrease in the mean of the self-reported pain scores in the first 24 hours using a Numerical visual scale

SECONDARY OUTCOMES:
decrease in pain on the EVN at 2 hours, 6 hours , Day 1 and Day 7 postoperative | 2 hours, 6 hours, Day 1 and Day 7 postoperative
  decrease in pain on the EVN at 2 hours, 6 hours , Day 1 and Day 7 with the pudental block method

CONTACTS AND LOCATIONS:
Locations (1):
- Camby, Montreuil, France

IPD SHARING:
Plan to Share IPD: No